CLINICAL TRIAL: NCT01742117
Title: Tailored Antiplatelet Initiation to Lesson Outcomes Due to Decreased Clopidogrel Response After Percutaneous Coronary Intervention (TAILOR-PCI)
Brief Title: Tailored Antiplatelet Therapy Following PCI
Acronym: TAILOR-PCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Spartan Bioscience Inc. (Industry); Applied Health Research Centre (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Naveen L. Pereira, Professor of Medicine, College of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-006837; 5U01HL128606 (NIH); 3U01HL128606-03S1 (NIH)
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Results first posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome; Stenosis
Keywords: percutaneous coronary intervention; angioplasty
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Constriction, Pathologic | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Genotype-Guided Therapy (Experimental): Subjects will be genotyped prospectively for CYP2C19*2, *3 and *17 alleles and will receive treatment based on their genotype. In this group, patients who have the CYP2C19 reduced function allele [i.e., *2 allele (heterozygous or homozygous) or *3 allele (heterozygous or homozygous)] patients will receive ticagrelor 90 mg bid. The WT YP2C19 patients will receive clopidogrel 75 mg once daily.
  Interventions: Drug: Clopidogrel; Drug: Ticagrelor
- Conventional Therapy (Active Comparator): Subjects will receive clopidogrel once daily after the index PCI and will be retrospectively genotyped for CYP2C19*2, *3 and *17 alleles after completion of one year of treatment with clopidogrel.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — One 75 mg tablet per day by mouth for one year
  Other Names: Plavix
Drug: Ticagrelor — One 90 mg tablet twice per day by mouth for one year
  Other Names: Brilinta
  Arms: Genotype-Guided Therapy

SUMMARY:
Clopidogrel is an anti-platelet medication approved by the U.S. Federal Drug Administration (FDA) for use in patients who undergo Percutaneous Coronary Intervention (PCI) with coronary stent implantation. Anti-platelet medications work to prevent blood clots from forming. Some studies have suggested that patients who have a certain genetic liver enzyme abnormality (known as cytochrome P450 2C19 [CYP2C19] *2 or *3 allele) may have a reduced ability to activate clopidogrel, and therefore may have a lowered response to clopidogrel. It is thought that perhaps people who have a coronary stent procedure may have this genetic liver enzyme abnormality. There is a research genetic test available to determine whether or not someone has this genetic liver enzyme abnormality. Ticagrelor, is a newer anti-platelet drug that is not dependent on the CYP2C19 liver enzyme for its activation and hence in poor clopidogrel metabolizers, alternative drugs like Ticagrelor have been recommended for use as an anti-platelet agent after PCI. The purpose of this study is to determine if genetic testing can identify the best anti-platelet therapy, for patients who undergo a coronary stent placement and do not activate clopidogrel very well.

DETAILED DESCRIPTION:
TAILOR-PCI is a multi-site, open label, prospective, randomized trial testing the hypothesis that after percutaneous coronary intervention (PCI), using a genotyping strategy ticagrelor 90 mg twice per day is superior to clopidogrel 75 mg per day in reducing a composite endpoint of major adverse cardiovascular events (MACE), i.e., non-fatal myocardial infarction, non-fatal stroke, severe recurrent ischemia, cardiovascular (CV) death, and stent thrombosis (primary endpoints) in CYP2C19 reduced function allele patients. Patients who undergo PCI will be randomized to a conventional therapy arm (i.e., to receive clopidogrel 75 mg once daily without prospective genotyping guidance) versus a prospective CYP2C19 genotype-based anti-platelet therapy approach (ticagrelor 90 mg bid in CYP2C19 *2 or *3 reduced function allele patients, clopidogrel 75 mg once daily in non-*2 or -*3 CYP2C19 patients). Buccal swabs will be obtained for those subjects randomized to the prospective genotyping arm. All subjects will have a blood sample drawn for DNA analysis but genotyping using these DNA samples will be performed only after completion of the duration of anti-platelet therapy (i.e., after one year). The primary endpoints will be assessed prospectively and will be compared between the conventional arm and the prospective genotyping arm among those identified as reduced function CYP2C19 allele carriers according to the 1-year genotype results.

ELIGIBILITY:
Inclusion

* Patient >18 years of age
* Patient presents with acute coronary syndrome (ACS) or stable coronary artery disease (CAD)
* Patient is eligible for PCI
* Patient is willing and able to provide informed written consent

5.3 Exclusion

* Patient not able to receive 12 months of dual anti-platelet therapy
* Failure of index PCI
* Patient or physician refusal to enroll in the study
* Patient with known CYP2C19 genotype prior to randomization
* Planned revascularization of any vessel within 30 days post-index procedure and/or of the target vessel(s) within 12 months post-procedure
* Anticipated discontinuation of clopidogrel or ticagrelor within the 12 month follow up period, example for elective surgery
* Serum creatinine >2.5 mg/dL within 7 days of index procedure
* Platelet count <80,000 or >700,000 cells/mm3, or white blood cell count <3,000 cells/mm3 if persistent (at least 2 abnormal values) within 7 days prior to index procedure.
* History of intracranial hemorrhage
* Known hypersensitivity to clopidogrel or ticagrelor or any of its components
* Patient is participating in an investigational drug or device clinical trial that has not reached its primary endpoint
* Patient previously enrolled in this study
* Patient is pregnant, lactating, or planning to become pregnant within 12 months
* Patient has received an organ transplant or is on a waiting list for an organ transplant
* Patient is receiving or scheduled to receive chemotherapy within 30 days before or after the procedure
* Patient is receiving immunosuppressive therapy or has known immunosuppressive or autoimmune disease (e.g., human immunodeficiency virus, systemic lupus erythematous, etc.)
* Patient is receiving chronic oral anticoagulation therapy (i.e., vitamin K antagonist, direct thrombin inhibitor, Factor Xa inhibitor)
* Concomitant use of simvastatin/lovastatin > 40 mg qd
* Concomitant use of potent CYP3A4 inhibitors (atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin and voriconazole) or inducers (carbamazepine, dexamethasone, phenobarbital, phenytoin, rifampin, and rifapentine)
* Non-cardiac condition limiting life expectancy to less than one year, per physician judgment (e.g. cancer)
* Known history of severe hepatic impairment
* Patient has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Patient has an active pathological bleeding, such as active gastrointestinal (GI) bleeding
* Inability to take aspirin at a dosage of 100 mg or less
* Current substance abuse (e.g., alcohol, cocaine, heroin, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5276 (Actual)
Dates: Start 2013-05; Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Pereira, MD, Principal Investigator — Mayo Clinic; Michael E Farkouh, MD, Principal Investigator — Toronto General Hospital; Kent R Bailey, PhD, Principal Investigator — Mayo Clinic
Locations (41):
- United States (26):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Sharp HealthCare, San Diego, California
  - Zuckerberg San Francisco General, San Francisco, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - NCH Heart Institute, Naples, Florida
  - NorthShore University Health System, Evanston, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - St. Elizabeth Healthcare, Crestview Hills, Kentucky
  - Henry Ford Hospital, Detroit, Michigan
  - Essentia Institute of Rural Health, Duluth, Minnesota
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - The University of Mississippi Medical Center, Jackson, Mississippi
  - Albany Medical College, Albany, New York
  - The Feinstein Institute for Medical Research, Manhasset, New York
  - Winthrop University Hospital, Mineola, New York
  - New York University Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Cardiology Associates of Schenectady, Schenectady, New York
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Greenville Health System, Greenville, South Carolina
  - MHS, Eau Claire, Eau Claire, Wisconsin
  - Mayo Clinic Health System, La Crosse, Wisconsin
  - Aurora Health Care, Milwaukee, Wisconsin
- Canada (8):
  - Vancouver General Hospital, UBC Division of Cardiology, Vancouver, British Columbia
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Humber River Hospital, Toronto, Ontario
  - Sunnybrook Health Services Center, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital - UHN, Toronto, Ontario
  - Regina General Hospital, Regina, Saskatchawan
- Mexico (3):
  - Hospital de Especialidades, Centro Medico Nacional 'La Raza', Mexico City
  - Hospital REgional No. 1, Mexico City
  - Hospital de Cardiologia, Centro Medico Nacional Siglo XXI, Mexico City
- South Korea (4):
  - Konyang University College of Medicine, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Ajou University Hospital, Gyeonggi-do
  - Chung-Ang University Hospital, Seoul

REFERENCES:
- [Result] Pereira NL, Farkouh ME, So D, Lennon R, Geller N, Mathew V, Bell M, Bae JH, Jeong MH, Chavez I, Gordon P, Abbott JD, Cagin C, Baudhuin L, Fu YP, Goodman SG, Hasan A, Iturriaga E, Lerman A, Sidhu M, Tanguay JF, Wang L, Weinshilboum R, Welsh R, Rosenberg Y, Bailey K, Rihal C. Effect of Genotype-Guided Oral P2Y12 Inhibitor Selection vs Conventional Clopidogrel Therapy on Ischemic Outcomes After Percutaneous Coronary Intervention: The TAILOR-PCI Randomized Clinical Trial. JAMA. 2020 Aug 25;324(8):761-771. doi: 10.1001/jama.2020.12443. PMID 32840598
- [Derived] Ingraham BS, Farkouh ME, Lennon RJ, So D, Goodman SG, Geller N, Bae JH, Jeong MH, Baudhuin LM, Mathew V, Bell MR, Lerman A, Fu YP, Hasan A, Iturriaga E, Tanguay JF, Welsh RC, Rosenberg Y, Bailey K, Rihal C, Pereira NL. Genetic-Guided Oral P2Y12 Inhibitor Selection and Cumulative Ischemic Events After Percutaneous Coronary Intervention. JACC Cardiovasc Interv. 2023 Apr 10;16(7):816-825. doi: 10.1016/j.jcin.2023.01.356. PMID 37045502
- [Derived] Mathew RO, Sidhu MS, Rihal CS, Lennon R, El-Hajjar M, Yager N, Lyubarova R, Abdul-Nour K, Weitz S, O'Cochlain DF, Murthy V, Levisay J, Marzo K, Graham J, Dzavik V, So D, Goodman S, Rosenberg YD, Pereira N, Farkouh ME. Safety and Efficacy of CYP2C19 Genotype-Guided Escalation of P2Y12 Inhibitor Therapy After Percutaneous Coronary Intervention in Chronic Kidney Disease: a Post Hoc Analysis of the TAILOR-PCI Study. Cardiovasc Drugs Ther. 2024 Jun;38(3):447-457. doi: 10.1007/s10557-022-07392-2. Epub 2022 Nov 29. PMID 36445624
- [Derived] Avram R, So D, Iturriaga E, Byrne J, Lennon R, Murthy V, Geller N, Goodman S, Rihal C, Rosenberg Y, Bailey K, Farkouh M, Bell M, Cagin C, Chavez I, El-Hajjar M, Ginete W, Lerman A, Levisay J, Marzo K, Nazif T, Olgin J, Pereira N. Patient Onboarding and Engagement to Build a Digital Study After Enrollment in a Clinical Trial (TAILOR-PCI Digital Study): Intervention Study. JMIR Form Res. 2022 Jun 13;6(6):e34080. doi: 10.2196/34080. PMID 35699977
- [Derived] Madan M, Abbott JD, Lennon R, So DYF, MacDougall AM, McLaughlin MA, Murthy V, Saw J, Rihal C, Farkouh ME, Pereira NL, Goodman SG; TAILOR-PCI Investigators *. Sex-Specific Differences in Clinical Outcomes After Percutaneous Coronary Intervention: Insights from the TAILOR-PCI Trial. J Am Heart Assoc. 2022 Jun 21;11(12):e024709. doi: 10.1161/JAHA.121.024709. Epub 2022 Jun 14. PMID 35699175
- [Derived] Baudhuin LM, Train LJ, Goodman SG, Lane GE, Lennon RJ, Mathew V, Murthy V, Nazif TM, So DYF, Sweeney JP, Wu AHB, Rihal CS, Farkouh ME, Pereira NL. Point of care CYP2C19 genotyping after percutaneous coronary intervention. Pharmacogenomics J. 2022 Dec;22(5-6):303-307. doi: 10.1038/s41397-022-00278-4. Epub 2022 Apr 21. PMID 35449399
- [Derived] Capodanno D, Angiolillo DJ, Lennon RJ, Goodman SG, Kim SW, O'Cochlain F, So DY, Sweeney J, Rihal CS, Farkouh M, Pereira NL. ABCD-GENE Score and Clinical Outcomes Following Percutaneous Coronary Intervention: Insights from the TAILOR-PCI Trial. J Am Heart Assoc. 2022 Feb 15;11(4):e024156. doi: 10.1161/JAHA.121.024156. Epub 2022 Feb 8. PMID 35132875
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Genotype-Guided Therapy | Conventional Therapy
Started | 2641 | 2635
Completed | 2641 | 2635
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Genotype-Guided Therapy | Conventional Therapy | Total
Number analyzed (Participants) | 2641 | 2635 | 5276
Age, Continuous [Median (Full Range); unit: years] | 62 [26 to 95] | 62 [21 to 93] | 62 [21 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 648 | 645 | 1293
  Male | 1993 | 1990 | 3983
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1750 | 1754 | 3504
  East Asian | 595 | 592 | 1187
  South Asian | 116 | 120 | 236
  African America | 57 | 67 | 124
  Other, Unknown or Not Reported | 123 | 102 | 225
  Hispanic or Latinx ethnicity | 78 | 70 | 148
Region of Enrollment [Number; unit: participants]
  Canada | 577 | 580 | 1157
  South Korea | 654 | 650 | 1304
  United States | 1359 | 1358 | 2717
  Mexico | 51 | 47 | 98

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of the a Major Adverse Cardiovascular Event in Subjects Identified as CPY2C19 LOF Carriers by TaqMan.
Description: Number of subjects who experienced major adverse cardiovascular event as defined as cardiovascular death, myocardial infarction, stroke, severe recurrent ischemia, and stent thrombosis in subjects identified as CPY2C19 LOF carriers by TaqMan.
Time Frame: 1 year after percutaneous coronary intervention (PCI)
Population: For 1 year endpoint in Genotype-Guided Therapy arm 1738 were excluded from data analysis due Identified as CYP2C19 LOF noncarriers by TaqMan or no TaqMan results available. For 1 year endpoint in Conventional Therapy arm 1689 were excluded from data analysis due Identified as CYP2C19 LOF noncarriers by TaqMan or no TaqMan results available.
Measure: Count of Participants; unit: Participants
Arm/Group | Genotype-Guided Therapy | Conventional Therapy
Number analyzed (Participants) | 903 | 946
Participants | 35 | 54

2. Secondary Outcome: Thrombolysis in Myocardial Infarction Major or Minor Bleeding in Subjects Identified as CPY2C19 LOF Carriers by TaqMan.
Description: Number of subjects that experienced thrombolysis in myocardial infarction major or minor bleeding in subjects identified as CYP2C19 LOF carriers by TaqMan
Time Frame: 1 year after percutaneous coronary intervention (PCI)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Genotype-Guided Therapy | Conventional Therapy
Number analyzed (Participants) | 903 | 946
Participants | 16 | 14

3. Secondary Outcome: Thrombolysis in Myocardial Infarction Major or Minor Bleeding
Description: Number of subjects that experienced thrombolysis in myocardial infarction major or minor bleeding
Time Frame: Approximately 3 years after percutaneous coronary intervention (PCI)
Measure: Count of Participants; unit: Participants
Arm/Group | Genotype-Guided Therapy | Conventional Therapy
Number analyzed (Participants) | 2641 | 2635
Participants | 54 | 53

4. Primary Outcome: Occurrence of the a Major Adverse Cardiovascular Event
Description: Number of subjects to experience a major adverse cardiovascular event as defined as cardiovascular death, myocardial infarction, stroke, severe recurrent ischemia, and stent thrombosis.
Time Frame: Approximately 3 years after percutaneous coronary intervention (PCI)
Measure: Count of Participants; unit: Participants
Arm/Group | Genotype-Guided Therapy | Conventional Therapy
Number analyzed (Participants) | 2641 | 2635
Participants | 262 | 269

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately one year on all participants.
Arm/Group | Genotype-Guided Therapy | Conventional Therapy
All-Cause Mortality (participants affected / at risk) | 95/2641 | 98/2635
Serious Adverse Events (participants affected / at risk) | 0/2641 | 0/2635
Other Adverse Events (participants affected / at risk) | 0/2641 | 0/2635

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT01742117/Prot_SAP_000.pdf